CLINICAL TRIAL: NCT03465475
Title: Anesthetic Cost Analysis With Desflurane in Automated Gas Control Mode With Maquet Flow-i Anaesthesia Machine
Brief Title: Anesthetic Cost Analysis With Desflurane in Automated Gas Control Mode
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yusuf Ziya ÇOLAK, Assistant Professor, Inonu University
Other Study IDs: Inonu uni
Record Dates: First submitted 2018-02-01; First posted 2018-03-14 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Safety Issues
Keywords: Low flow anesthesia; Desflurane; Cost analysis; Automated gas control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: The patient who receive 300 mL fresh gas flow with AGC mode during the general anesthesia
- Group 2: The patient who receive 600 mL fresh gas flow with AGC mode during the general anesthesia
- Group 3: The patient who receive 600 mL fresh gas flow with manuelly during the general anesthesia

SUMMARY:
Inhalation agents constitute the major part of anesthetic drug costs (20% - 25%) and a significant portion of the applied inhalation agents are thrown into the atmosphere through the waste gas system without being absorbed by the patient. The amount of waste gas is directly correlated to the fresh gas flow (FGF). Reducing the TGA during general anesthesia reduces the consumption of inhalant agents and contributes to the reduction of greenhouse gas pollution. Risks such as hypoxia, hypercapnia, inadequate depth of anesthesia and potential toxic gas accumulation were associated with low flow anesthesia, but the patient was provided with adequate safety by following pulse oximetry, capnography, FiO2 and anesthetic gas analysis. We aimed to perform anesthetic cost analysis and patient security in automated gas control mode (AGC).

DETAILED DESCRIPTION:
After the ethical approvel 60 adult patients scheduled for hepatectomy will be taken to study. Patients will be monitored after they are taken to the operating room (ECG, NIBP, SpO2, Body Temp, BIS, NIRS, PVI, PI, ORI). After the anesthesia induction and tarakeal entubation, first twenty patient will take 300 mL fresh gas flow with AGC mode (group 1), Second twenty patient will take 600 mL fresh gas flow with AGC mode (group 2), third twenty patient will take 600 mL fresh gas flow with manually. Hemodynamic and gas consumption data will be recorded. An operating room will be reserved for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing hepatectomy with general anesthesia

Exclusion Criteria:

* Essential data missing
* Patient participating in other research projects
* Drug allergy
* Anesthetic complication story

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hepatectomy operation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Amount of used anesthetic gas (desflurane) | Through study completion, an average of 2 month
  Amount of used desflurane will be determined in milliliter by anesthesia machine (Maquet Flow i40) for each patient.

SECONDARY OUTCOMES:
Heart rate | Through study completion, an average of 2 month
  Heart rate/min
Mean arterial pressure | Through study completion, an average of 2 month
  Mean arterial pressure (mm/Hg)
Peripheral oxygen saturation | Through study completion, an average of 2 month
  Peripheral oxygen saturation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Z Çolak, MD, Principal Investigator — Investigator
Locations (1):
- Inonu Univercity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No